CLINICAL TRIAL: NCT01333618
Title: Introducer Curving Technique for Tilt of Transfemoral Günther Tulip Inferior Vena Cava Filter：A Randomized Double-Blind Comparison
Brief Title: Introducer Curving Technique for Tilt of Transfemoral Günther Tulip Inferior Vena Cava Filter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University, China (Other)
Responsible Party: Liang Xiao Associate professor, Department of Radiology, the First Hospital of China Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: LXiao-01
Record Dates: First submitted 2011-04-04; First posted 2011-04-12 (Estimated); Last update posted 2011-04-26 (Estimated); Status verified 2008-08

CONDITIONS: Deep Venous Thrombosis
Keywords: Filter Tilt; Preventional efficiency; Günther Tulip filter; Transfemoral Approach
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- curving introducer (Experimental)
  Interventions: Device: curving introducer Günther Tulip Filter
- straight introducer (Placebo Comparator)
  Interventions: Device: straight introducer Günther Tulip Filter

INTERVENTIONS:
Device: curving introducer Günther Tulip Filter — The Günther Tulip filter (Vena Cava MReye Filter Set; William Cook Europe, Bjaeverskov, Denmark) The amplitude of introducer curvature was 5°-15° less than the angle between the inferior vena cave axis and the approached iliac vein axis and the distance between the vertex of the curved angle and the hook of the filter was 2-4cm less than the distance between the level of the renal vein confluence and the furcation of inferior vena cave.
  Arms: curving introducer
Device: straight introducer Günther Tulip Filter — The Günther Tulip filter (Vena Cava MReye Filter Set; William Cook Europe, Bjaeverskov, Denmark)
  Arms: straight introducer

SUMMARY:
It has been demonstrated that implantation of inferior vena cava filter was safe and effective in the prevention or reduction of fatal pulmonary thromboembolism in numerous clinical researches. When acute deep venous thrombosis need transcatheter thrombolysis, transfemoral Günther Tulip Filter implantation could avoid catheter across the Günther Tulip Filter. Although incidence of significant filter tilting (>10°) is not high (13%-16%), severe tilting of the Günther Tulip Filter may be associated with difficulty or sometimes impossibility of retrieval. It has been reported that a simple technique of keeping tension of the delivery system may prevent significant tilting of the transjugular Günther Tulip Filter in an in-vitro study. But no clinical study of prevention transfemoral Günther Tulip Filter from tilting has been reported. The investigators conducted a randomized, controlled study to test whether the introducer curving technique is useful to decrease the extent of tilting of transfemoral Günther Tulip Filter.

DETAILED DESCRIPTION:
The study was designed as a double-blind randomized controlled trial, with research assessors and patients intended to be blind to the intervention status. The staff members performing the assessment were not involved in implementing any aspect of the intervention. 108 patients were randomized to accept curving introducer Günther Tulip Filter and transcatheter thrombolysis or straight introducer Günther Tulip Filter and transcatheter thrombolysis. The assessments include the tilting angle between the axes of inferior vena cava and Günther Tulip Filter after implantation; the tilting angle between the axes of inferior vena cava and Günther Tulip Filter before retrieval; the fluoroscopy time of Günther Tulip Filter retrieval; the rate of retrieval hook adhering vascular wall; the success rate of retrieval.

ELIGIBILITY:
Inclusion Criteria:

* acute lower extremity deep vein thrombosis, diagnosed by vascular ultrasound and clinical history

Exclusion Criteria:

* both lower extremities deep vein thrombosis
* Inferior Vena Cava thrombosis
* refractory hypertension (blood pressure > 180/110mmHg)
* contraindication of thrombolysis
* the diameter of Inferior Vena Cava > 35mm or < 14mm
* Inferior Vena Cava venous anomalies

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2008-09; Primary Completion 2010-06 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
the tilting angle between the axes of Inferior Vena Cava and Günther Tulip Filter after implantation | just after filter implantation （up to 24 hours）

SECONDARY OUTCOMES:
the tilting angle between the axes of Inferior Vena Cava and Günther Tulip Filter before retrieval | just before filter retrieval （up to 90 days）
the fluoroscopy time of Günther Tulip Filter retrieval | just after filter retrieval（up to 90 days）
the rate of retrieval hook adhering vascular wall | just after filter retrieval（up to 90 days）
the success rate of retrieval | just after filter retrieval（up to 90 days）

CONTACTS AND LOCATIONS:
Overall Officials: Liang Xiao, Ph.D. M.D., Study Director — First Hospital of China Medical University
Locations (1):
- Department of Radiology, the First Hospital of China Medical University, Shenyang, Liaoning, China